CLINICAL TRIAL: NCT06054555
Title: A Randomized, Double-Blind Study Evaluating the Efficacy, Safety, and Immunogenicity of ABP 206 Compared With OPDIVO® (Nivolumab) in Subjects With Treatment-Naïve Unresectable or Metastatic Melanoma
Brief Title: A Study to Evaluate ABP 206 Compared With OPDIVO® (Nivolumab) in Subjects With Unresectable or Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210031; 2023-503288-40 (EudraCT Number)
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
Keywords: Treatment-naive; Unresectable melanoma; Metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study is double-blinded; therefore, the investigators, study personnel (with the exception of the data monitoring committee, authorized unblinded sponsor and contract research organization staff, and unblinded site pharmacy staff) and the study subjects will remain blinded to treatment allocation. ABP 206 and nivolumab will be coded and labeled to protect blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABP 206 (Experimental): Subjects will receive Dose A of ABP 206 via intravenous (IV) infusion.
  Interventions: Drug: ABP 206
- Nivolumab (Active Comparator): Subjects will receive Dose A of Nivolumab via IV infusion.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: ABP 206 — ABP 206 will be given intravenously over a period of 30 or 60 minutes, every 4 weeks (Q4W) for a total of 24 months.
  Arms: ABP 206
Drug: Nivolumab — Nivolumab will be given intravenously over a period of 30 or 60 minutes, Q4W for a total of 24 months.
  Other Names: OPDIVO®
  Arms: Nivolumab

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and immunogenicity of ABP 206 compared with Nivolumab in Subjects with Treatment-Naïve Unresectable or Metastatic Melanoma.

DETAILED DESCRIPTION:
Eligible subjects will be randomized (1:1) to receive investigational product (ABP 206 or nivolumab).

All subjects will be treated until disease progression, unacceptable toxicity, or subject withdrawal of consent for a maximum of 24 months of treatment.

The total duration of study participation for each subject will be approximately 26 months.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 18 years of age.
* Histologically confirmed unresectable or metastatic melanoma.
* Subject has no prior systemic treatment for advanced disease.
* Subject must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
* Tumor tissue from site of unresectable or metastatic melanoma must be available for biomarker analyses in order to be randomized.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.

Key Exclusion Criteria:

* Subject has had any prior systemic anti-cancer therapy for the treatment of advanced melanoma.
* Known hypersensitivity to monoclonal antibodies or to any of the excipients of the study drug.
* Subject has active central nervous system (CNS) metastases not previously treated.
* Ocular melanoma.
* Subject has active or known immune-mediated disorders.
* Subject has had prior treatment with PD-1/PD-L1 and cytotoxic T lymphocyte- associated protein 4 inhibitors, or other antibodies targeting immune checkpoint pathways.
* Subject has medical conditions requiring systemic immunosuppression with either corticosteroids or other immunosuppressive medications within 14 days of the first dose of investigational product.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2028-01-25 (Estimated); Study Completion 2028-01-25 (Estimated)

PRIMARY OUTCOMES:
Objective response by Week 49 | Week 49
Objective response at Week 17 | Week 17
Progression-free survival (PFS) | From Randomization until Follow-up or End of treatment (EOT) or Early termination (ET) (Approximately 105 Weeks)
Overall survival (OS) | From Randomization until Follow-up or EOT or ET (Approximately 105 Weeks)
Duration of response (DOR) | From Randomization until Follow-up or EOT or ET (Approximately 105 Weeks)

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events | Week 1 until Week 105
Number of subjects with treatment-emergent serious adverse events | Week 1 until Week 105
Number of subjects with treatment-emergent adverse events of interest | Week 1 until Week 105
Number of subjects with anti-drug antibodies | Predose on Week 1 (Baseline), Weeks 9, 17, 29, 41, 53, 65, 77, 89, 101 and Week 105
Serum concentrations of ABP 206 and nivolumab (Ctrough) | Predose on Week 1 (Baseline), Weeks 9, 17, 29, 41, 53, 65, 77, 89, 101 and Week 105

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (180):
- United States (5):
  - Cancer and Blood Specialty clinic, Long Beach, California
  - Fort Wayne Medical Oncology and Hematology - Office of Clinical Research, Fort Wayne, Indiana
  - Our Lady of the Lake Physicians Group-Medical Oncology-Woman's Pavilion, Baton Rouge, Louisiana
  - Oncology Hematology Associates, Springfield, Missouri
  - Hematology-Oncology Associates of Central New York, P.C. (HOA) - East Syracuse - CCOP, East Syracuse, New York
- Argentina (5):
  - Centro de Investigaciones Médicas y Desarrollo LC, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Centro De Investigaciones Medicas Mar Del Plata (CIMMDP) - Rheumatology, Mar Del Plata, Río Negro Province
  - Clínica Viedma - Oncology, Viedma, Río Negro Province
  - Instituto De Oncologia De Rosario, Rosario, Santa Fe Province
  - ISIS Clinica Especializada, Santa Fe
- Bosnia and Herzegovina (4):
  - Clinical Center University of Sarajevo - Clinic of Oncology, Sarajevo, Kanton Sarajevo
  - University Clinical Center of Republic of Srpska, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla - Oncology, Hematology and Radio, Tuzla, Tuzlanski Kanton
  - Cantonal hospital Zenica - Oncology, Zenica, Zeničko-dobojski Kanton
- Dr. Everett Chalmers Hospital - Oncology, Fredericton, New Brunswick, Canada
- Chile (4):
  - IC La Serena Research, La Serena, Coquimbo Region
  - Centro de Investigacion y Desarrollo Oncologico, Temuco, Región de la Araucanía
  - Oncocentro Apys, Valparaíso, Región de Valparaíso
  - Icegclinic Research & Care, Estacion Central, Santiago Metropolitan
- Croatia (3):
  - University Hospital Centre Zagreb - Oncology department, Zagreb, City of Zagreb
  - Poliklinika Anova, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek, Osijek, Osjecko-baranjska Županija
- Czechia (2):
  - FN Hradec Kralove - Klinika onkologie a radioterap, Hradec Kralove, Moravskoslezský kraj
  - Vseobecna fakultni nemocnice v Praze - Dermatovenerologicka, Prague
- Tartu University Hospital - Oncology, Tartu, Tartu, Estonia
- France (3):
  - CHU de Poitiers, Poitier, Haute-Vienne
  - Centre Hospitalier De Saint Malo - Oncologie, Rennes, Ille-et-Vilaine
  - C.H.R.U Hopital Claude Huriez - Dermatologie, Lille, Nord
- Georgia (5):
  - LTD "High technology hospital MEDCENTER", Batumi, Adjara
  - LLC "Todua Clinic", Tbilisi
  - LTD "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi
  - JSC "K.Eristavi National Center of Experimental and Clinical Surgery", Tbilisi
  - LTD "Multprofile Clinic Consilium Medulla" - Oncology, Tbilisi
- Germany (3):
  - Goethe University Frankfurt, Frankfurt am Main, Hesse
  - Philipps-University Marburg, Marburg, Hesse
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
- Italy (22):
  - Ospedale Maggiore Di Crema - Oncologia e Day Hospital oncologico, Crema, Cremona
  - IRST Dino Amadori (IRST IRCCS) - UNK, Meldola, Forli
  - PO Ospedale San Vincenzo - Oncologia Medica, Taormina, Messina
  - Istituto Clinico Humanitas, Rozzano, Milano
  - AO Ss Antonio, Biagio e Arrigo, Alessandria
  - AUO Consorziale-Policlinico Bari, Bari
  - Istituto dei Tumori Giovanni Paolo II - Oncologia Medica - Tumori Rari e Melanoma, Bari
  - ASST Papa Giovanni XXIII - Oncologia, Bergamo
  - AOU Careggi, Florence
  - IRCCS Ca'Granda Maggiore Policlinic, Milan
  - Ospedale San Raffaele, IRCCS - Oncologia Medica, Milan
  - AOU Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Sanitaria Locale Napoli 1 Centro (ASL Napoli 1) - Ospedale del Mare, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario Campus Bio-medico - Oncologia Medica, Roma
  - IRCCS IFO, Istituto Nazionale dei Tumori Regina Elena (IRE), Roma
  - Istituto Dermopatico dell'Immacolata (IDI) - IRCCS - Oncologia, Roma
  - Ospedale Isola Tiberina - Gemelli Isola - Oncologia Medica, Roma
  - AOU Senese, Policlinico Le Scotte, Siena
  - Ospedale di Circolo, Presidio di Varese - Oncologia, Varese
- Jordan (4):
  - Al Khalidi Hospital and Medical Center - Research, Amman, 'Ammān
  - The Speciality Hospital (TSH) / Advanced Clinical Center, Amman, 'Ammān
  - King Hussein Cancer Center, Amman
  - Pharmaceutical Research Center (KAUH), Irbid
- Lebanon (6):
  - Saint George Hospital University Medical Center, El Achrafiyé, Beyrouth
  - Nini Hospital, Tripoli, Loubnâne Ech Chemâli
  - Hammoud Hospital University Medical Center (HHUMC) - Hemato-Oncology, Saida, Loubnâne Ej Jnoûbi
  - Ain Wazein Hospital - internal medicine, Beirut
  - American University of Beirut Medical Center - Haematology, Beirut
  - Hotel Dieu de France Hospital - Oncology, Beirut
- National Cancer Institute - Conservative Tumour Therapy, Vilnius, Vilnius County, Lithuania
- Malaysia (7):
  - Hospital Pulau Pinang, Pulau Pinang, Pahang
  - Sarawak General Hospital, Kuching, Sarawak
  - National Cancer Institute - Radiotherapy and Oncology, Putrajaya, Selangor
  - HOSPITAL UNIVERSITI SAINS MALAYSIA - Pediatrics, Kubang Kerian, Terengganu
  - Hospital Kuala Lumpur - Surgery, Kuala Lumpur, Wilayah Persekutuan Kuala Lump
  - Hospital Canselor Tuanku Muhriz UKM, Kuala Lumpur, Wilayah Persekutuan Kuala Lump
  - Pantai Hospital Kuala Lumpur - Oncology, Kuala Lumpur, Wilayah Persekutuan Kuala Lump
- Mexico (15):
  - Preparaciones Oncologica SC, León, Guanajuato
  - Centro de Inm Onc de Occ Sa de Cv, Guadalajra, Jalisco
  - Health Pharma Professional Research S.A de C.V., Mexico City, Mexico City
  - iCan Oncology Center Centro Medico AVE, Monterrey, Nuevo León
  - Centro Medico Zambrano Hellion TecSalud, Monterrey, Nuevo León
  - Althian - Research Management Center, San Pedro Garza García, Nuevo León
  - Centro de Estudios y Prevención del Cancer AC, Juchitán de Zaragoza, Oaxaca
  - Hospital Angeles Centro Médico San Luis Potosí - Cardiologia, San Luis Potosí City, San Luis Potosí
  - Neurosciences Hospital Angeles Culiacán - Neurociencias Estudios Clínicos S.C., Culiacán, Sinaloa
  - Centro de Atención e Investigación Clínica en Oncología, Mérida, Yucatán
  - Centro de Investigación Médica Aguascalientes (CIMA) - Oncology, Aguascalientes
  - Boca Clinical Trials MÃ©xico, Guadalajara
  - Oncare Cancer Center Viaducto CdMx, Mexico City
  - ONCOCENTER PUEBLA - Dermatology, Puebla City
  - Clinical Research Institute, Tlalnepantla
- Arensia Exploratory Medicine - Moldova - IMSP Institutul Oncologic - Oncology, Chisinau, Moldova, Republic of, Moldova
- Amphia Ziekenhuis - Molengracht, Breda, North Brabant, Netherlands
- Philippines (9):
  - Baguio General Hospital and Medical Center - Oncology, Baguio City, Benguet
  - Cebu Doctors' University Hospital - Oncology, Cebu City, Cebu
  - The Medical City - Clinical Research Unit, Iloilo City, Iloilo
  - The Medical City - Neurology, Pasig, Metropolitan Manila
  - Cagayan de Oro Medical Center - Internal Medicine, Cagayan de Oro, Misamis Oriental
  - Center for Skin Research, Testing and Product Development, Makati City, National Capital Region
  - Philippine General Hospital, Manila/Ermita, National Capital Region
  - Cardinal Santos Madical Center, San Juan City, National Capital Region
  - Riverside Medical Center, Bacolod, Negros Occidental
- Portugal (6):
  - Centro Hospitalar de Setúbal - Oncologia, Setúbal, Setúbal District
  - Champalimaud Cancer Center, Lisbon
  - Unidade Local De Saude De Lisboa Ocidental E.P.E., Lisbon
  - Centro Hospitalar de Lisboa Norte E.P.E. - H. Santa Maria Serviço de Oncologia Médica, Lisbon
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil - Oncologia Medica, Lisbon
  - Instituto Português Oncologia Francisco Gentil do Porto - Oncologia Medica, Porto
- Romania (12):
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca - Medical Oncology, Cluj-Napoca, Cluj
  - Medisprof - Medical Oncology, Cluj-Napoca, Cluj
  - Radiotherapy Center Cluj - Medical Oncology, Floreşti, Cluj
  - Oncolab - Medical Oncology, Craiova, Dolj
  - Centrul de Oncologie Sf Nectarie - Medical Oncology, Craiova, Dolj
  - Medical Center Gral, Ploieşti, Prahova
  - Spitalul Municipal Ploiesti - Oncologie, Ploieşti, Prahova
  - Oncocenter- Oncologie Clinica - Medical Oncology, Timișoara, Timiș County
  - Memorial Healthcare International - Oncology, Bucharest
  - Institutul Oncologic Prof Dr Alexandru Trestioreanu Bucuresti - Medical Oncology I, Bucharest
  - Centrul de Oncologie Euroclinic - Oncology, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu - Oncologie, Sibiu
- Serbia (2):
  - Institute for Oncology of Vojvodina, Clinic for Internal Oncology-Department of Soft Tissue, Skin, B, Kamenitz, Vojvodina
  - University Clinical Center of Kragujevac, Center for Internal Oncology, Kragujevac, Šumadijski Okrug
- South Africa (9):
  - Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Wits Clinical Research, Parktown, Johannesburg, Gauteng
  - Steve Biko Academic Hospital, Pretoria, Gauteng
  - Curo Oncology, Pretoria, Gauteng
  - Little Company Of Mary Hospital - Oncology, Pretoria, Gauteng
  - Rainbow Oncology Centre, Durban, KwaZulu-Natal
  - Cape Gate Oncology Centre, Cape Town, Western Cape
  - Cancercare - Rondebosch Oncology, Cape Town, Western Cape
- South Korea (5):
  - Inje University Haeundae Paik Hospital - Oncology, Busan, Busan Gwang'yeogsi [Pusan-Kwan
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido [Kyonggi-do]
  - Severance Hospital, Yonsei University Health System - Division of Medical Oncology, Department of In, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Asan Medical Center - Oncology, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Samsung Medical Center - Family Medicine, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
- Spain (10):
  - Hospital Universitario Virgen de la Macarena - Oncología Médica, Seville, Andalusia
  - Institut Català d'Oncologia-Hospital Universitari Germans Trias i Pujol - Oncología Médica, Badalona, Barcelona
  - Hospital San Pedro de Alcántara - Oncología, Cáceres, Cáceres
  - H.U.V.Arrixaca - Oncología, El Palmar, Murcia, Región de
  - Hospital Universitario Vall d'Hebron - Oncología Médica, Barcelona
  - Hospital de la Santa Creu i Sant Pau - Oncología Médica, Barcelona
  - M.D. Anderson Center Madrid, Madrid
  - Hospital Regional Universitario de Malaga - Servicio de Oncología, Málaga
  - Hospital HLA Jerez Puerta Sur, Seville
  - Consorcio Hospital General Universitario de Valencia - Oncología, Valencia
- Taiwan (4):
  - China Medical University Hospital - Internal Medicine, Taichung, Taichung Municipality
  - Taipei Medical University - Shuang Ho Hospital Ministry of Health and Welfare, New Taipei City, Taipei
  - Changhua Christian Medical Foundation - Changhua Christian Hospital - Internal Medicine, Changhua
  - Taipei Municipal Wanfang Hospital - Managed by Taipei Medical University - Hematology and Oncology, Taipei
- Thailand (6):
  - Khon Kaen University, Srinagarind Hospital - Academic Clinical Research Office (ACRO), Khonkaen, Changwat Khon Kaen
  - Prince of Songkla University, Songkhla, Changwat Songkhla
  - Maharaj Nakorn Chiangmai Hospital - Medical Oncology, Muang, Chiang Mai
  - King Chulalongkorn Memorial Hospital [Medical Oncology], Bangkok, Krung Thep Maha Nakhon [Bangko
  - Siriraj Hospital - Medical Oncology, Bangkok, Krung Thep Maha Nakhon [Bangko
  - Ramathibodi Hospital - Immunology and Rheumatology, Rajthevi, Krung Thep Maha Nakhon [Bangko
- Turkey (Türkiye) (20):
  - Gazi University Medical Faculty - Gynecology, Yenimahalle/Ankara, Ankara
  - Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital - Medical Oncology, Kadıköy, Istanbul
  - Adana City Training and Research Hospital, Adana
  - Gulhane Training and Research Hospital - Medical Oncology, Ankara
  - Ankara University Medical Faculty - Medical Oncology, Ankara
  - Ankara Liv Hospital, Ankara
  - Memorial Ankara Hospital - Oncology, Ankara
  - Dr Abdurrahman Yurtaslan Training and Research Hospital - Medical Oncology, Ankara
  - Uludag University Medical Faculty, Bursa
  - Medical Point Gaziantep Hospital - Medical Oncology, Gaziantep
  - Gaziantep University Sahinbey Practise and Research Hospital - Internal Medicine- Endocrinology and, Gaziantep
  - BakirkÃ¶y Dr. Sadi Konuk EÄŸitim ve AraÅŸtirma Hastanesi - Oncology, Istanbul
  - Koc Universitesi Hastanesi; Tıbbi Onkoloji, Istanbul
  - Memorial Bahçelievler Hospital, Istanbul
  - Izmir Medical Point Hastanesi, Izmir
  - Kocaeli University Research and Practice Hospital - Medical Oncology, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty - Oncology, Konya
  - Sakarya Training and Research Hospital, Sakarya
  - VM Medical Park Samsun Hospital - Medical oncology, Samsun
  - Namik Kemal Universitesi - Tip Fakultesi, Tekirdağ
- TOV "ARENSIIa EKSPLORATORI MEDISIN", Kyiv, Kyïv, Ukraine
- Vietnam (3):
  - Hanoi Oncology Hospital, Hanoi, Ha Noi, Thu Do
  - Vietnam National Cancer Hopsital, Hanoi, Ha Noi, Thu Do
  - HCM Oncology Hospital - Medical Oncology, Ho Chi Minh City, Ho Chi Minh, Thanh Pho [Sai Go

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues, and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data-sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data-sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com